CLINICAL TRIAL: NCT04125901
Title: Chronic Idiopathic Neck Pain in High School Students: Effectiveness of an Intervention Based on Exercise and Pain Neuroscience Education
Brief Title: Pain Neuroscience Education and Exercise in High School Students With Chronic Idiopathic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aveiro University (Other)
Collaborators: Foundation for Science and Technology, Portugal (Other)
Responsible Party: Principal Investigator, Rosa Andias, Physiotherapist (Master), Aveiro University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24092019
Record Dates: First submitted 2019-10-01; First posted 2019-10-14 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Chronic Neck Pain
Keywords: Chronic Neck Pain; Adolescents; Pain Neuroscience Education; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Neuroscience Education and Exercise (Experimental): Participants will received an 8-week intervention consisting of exercise and pain neuroscience education. Pain neuroscience education will be conducted in line with international guidelines and will address the following topics: pain neurophysiology, nociception and nociceptive pathways, inhibition and spinal cord stimulation, peripheral and central sensitization, nervous system plasticity and the impact of variables such as stress, anxiety, sleep and exercise on pain behavior. Exercise will be performed in accordance with international guidelines for chronic NP. Motor control, endurance and strengthening exercises will be performed for the neck and scapulo-thoracic region.
  Interventions: Other: Pain Neuroscience Education and Exercise
- Exercise (Other): Participants will received an 8-week intervention consisting of exercise. The exercise performed in this group will be the same as in the intervention group and will follow the same international guidelines for chronic NP.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Pain Neuroscience Education and Exercise — The incorporation of the exercise in this group will be gradual, in order to decrease the education component and increase the exercise component (up to 45/60 minutes). The 1st session will be only PNE and will last approximately 45 minutes. In the 2nd session, there will be 30 minutes of PNE and the remaining 15 minutes of exercise. In the following 4th and 6th sessions, 15 minutes of each session will be used to clarify doubts and emphasize PNE concepts and strategies. The 8th session will include exercises only. In WhatsApp sessions, in addition to the video with the exercises, participants will receive activities about the PNE.
  Arms: Pain Neuroscience Education and Exercise
Other: Exercise — The exercise group will perform exercises in all sessions (45 minutes of exercise in face-to-face sessions). In WhatsApp sessions, participants will receive a video with exercises to perform at home.
  Arms: Exercise

SUMMARY:
Musculoskeletal pain can affect up to 40% of children and adolescents. Neck pain (NP) is one of the most prevalent painful conditions and evidence suggests that its prevalence has increased in recent decades in adolescents aged 16 to 18 years, from 22.9% in 1991 to 29.5% in 2011. Interventions based on pain neuroscience education have emerged as promising strategies in chronic pain conditions.In adults this intervention has been explored in many pain conditions, including musculoskeletal pain, but there is only one pilot study in adolescents with chronic NP and one case study in adolescents with fibromyalgia.

Thus, the main objective of the present study is:

(i) To compare the effectiveness of an education program based on pain neuroscience education and exercise versus exercise alone, in decreasing pain intensity in secondary school students with chronic and idiopathic NP immediately after the intervention and at 6 months.

The secondary objectives are to:

i) Compare the effectiveness of these programs immediately after the intervention and at 6 months in i) disability, ii) sleep, iii) pain catastrophizing, iv) fear of movement, v) self-efficacy, vi) central sensitization vii) the strength of the deep neck flexors and extensors muscles and stabilizers of the scapula; and viii) the pressure pain threshold between the two intervention groups;

ii) Explore possible predictors of response to treatment.

DETAILED DESCRIPTION:
It is anticipated that the sample will consist of 127 participants from four secondary schools that will be divided into two groups. Both groups will receive the same exercise-based intervention. The experimental group will receive, in addition to exercise, an intervention based on pain neuroscience education. The intervention will consist of 1 session per week during 8 weeks and will be applied in small groups.

The intervention will be performed in a blended-learning format. Five sessions will be face-to-face with up to 45 minutes duration, performed at school and incorporated into physical education classes and 3 will be performed at home, supported by vídeos sent by WhatsApp. The first two sessions will always be face-to-face. Face-to-face sessions will be interspersed with WhatsApp sessions.

Participants will be assessed, by online questionnaires, for sociodemographic aspects, pain characterization and physical activity level, disability, sleep, catastrophizing, fear of movement, self-efficacy, central sensitization and knowledge on pain neurophysiology. In addition, 3 muscle tests will be performed for the deep neck flexor and extensor muscles and scapular stabilizers, and the pressure pain thresholds in the neck and at distance will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Students with chronic and idiopathic NP for at least 3 months
* Have a pain intensity of NPS greater than or equal to 2
* Not receiving any treatment for NP (except analgesic)

Exclusion Criteria:

* All students with nervous or rheumatic system pathology
* Students attending special education (because they may need more accompaniment which, in this group intervention, will not be possible)

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Aged between 15 and 18 years
Enrollment: 127 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Intensity of pain | Baseline
  Assessed using the numeric rating scale that assesses pain intensity (range 0-10 and higher values are indicative of higher pain intensity)
Intensity of pain | 8 weeks
  Assessed using the numeric rating scale that assesses pain intensity (range 0-10 and higher values are indicative of higher pain intensity)
Intensity of pain | 6 months
  Assessed using the numeric rating scale that assesses pain intensity (range 0-10 and higher values are indicative of higher pain intensity)

SECONDARY OUTCOMES:
Pain location | Baseline
  Assessed using a body chart where the patients identifies the painful body segments
Pain location | 8 weeks
  Assessed using a body chart where the patients identifies the painful body segments
Pain location | 6 months
  Assessed using a body chart where the patients identifies the painful body segments
Pain frequency | Baseline
  Assessed using a closed question about pain frequency in the last week. (How many times in the last week have you felt this pain?". The answer options are: Never, rarely (once a week) occasionally (2 to 3 times a week), often (more than 3 times a week) and always.
Pain frequency | 8 weeks
  Assessed using a closed question about neck pain frequency in the last week (How many times in the last week have you felt this pain?". The answer options are: Never, rarely (once a week) occasionally (2 to 3 times a week), often (more than 3 times a week) and always.
Pain frequency | 6 months
  Assessed using a closed question about neck pain frequency in the last week (How many times in the last week have you felt this pain?". The answer options are: Never, rarely (once a week) occasionally (2 to 3 times a week), often (more than 3 times a week) and always.
Physical activity | Baseline
  Assessed using two questions regarding moderate or vigorous physical activity during the week ("In addition to your physical education classes, did you perform any other moderate physical activity?" and "In addition to your physical education classes, did you perform any other vigorous physical activity?") adapted by Silva et al. 2017.
Physical activity | 8 weeks
  Assessed using two questions regarding moderate or vigorous physical activity during the week ("In addition to your physical education classes, did you perform any other moderate physical activity?" and "In addition to your physical education classes, did you perform any other vigorous physical activity?") adapted by Silva et al. 2017.
Physical activity | 6 months
  Assessed using two questions regarding moderate or vigorous physical activity during the week ("In addition to your physical education classes, did you perform any other moderate physical activity?" and "In addition to your physical education classes, did you perform any other vigorous physical activity?") adapted by Silva et al. 2017.
Disability | Baseline
  Assessed using the Functional Disability Inventory (Total score range from 0-60 and higher scores are indicative of greater pain-related disability)
Disability | 8 weeks
  Assessed using the Functional Disability Inventory (Total score range from 0-60 and higher scores are indicative of greater pain-related disability)
Disability | 6 months
  Assessed using the Functional Disability Inventory (Total score range from 0-60 and higher scores are indicative of greater pain-related disability)
Sleep | Baseline
  Assessed using the Basic Scale of Symptoms of Insomnia and Sleep Quality (Total score range from 0-28 and higher scores are indicative of poorer sleep quality)
Sleep | 8 weeks
  Assessed using the Basic Scale of Symptoms of Insomnia and Sleep Quality (Total score range from 0-28 and higher scores are indicative of poorer sleep quality)
Sleep | 6 months
  Assessed using the Basic Scale of Symptoms of Insomnia and Sleep Quality (Total score range from 0-28 and higher scores are indicative of poorer sleep quality)
Pain catastrophizing | Baseline
  Assessed using the Pain Catastrophizing Scale (Total score range from 0-52 and higher values are indicative of higher pain catastrophizing)
Pain catastrophizing | 8 weeks
  Assessed using the Pain Catastrophizing Scale (Total score range from 0-52 and higher values are indicative of higher pain catastrophizing)
Pain catastrophizing | 6 months
  Assessed using the Pain Catastrophizing Scale (Total score range from 0-52 and higher values are indicative of higher pain catastrophizing)
Fear of movement | Baseline
  Assessed using the Tampa Scale of Kinesiophobia (Total score range from 13-52 and higher values are indicative of higher levels of fear of movement)
Fear of movement | 8 weeks
  Assessed using the Tampa Scale of Kinesiophobia (Total score range from 13-52 and higher values are indicative of higher levels of fear of movement)
Fear of movement | 6 months
  Assessed using the Tampa Scale of Kinesiophobia (Total score range from 13-52 and higher values are indicative of higher levels of fear of movement)
Self-efficacy | Baseline
  Assessed using the Self-Efficacy Pain Scale (Total score range from 7 to 35 points and lower scores are indicate of greater self-efficacy)
Self-efficacy | 8 weeks
  Assessed using the Self-Efficacy Pain Scale (Total score range from 7 to 35 points and lower scores are indicate of greater self-efficacy)
Self-efficacy | 6 months
  Assessed using the Self-Efficacy Pain Scale (Total score range from 7 to 35 points and lower scores are indicate of greater self-efficacy)
Central Sensitization | Baseline
  Assessed using the Central Sensitization Inventory (Total score range from 0 to 100 and higher scores are indicative of a higher degree of symptomatology associated with central sensitization)
Central Sensitization | 8 weeks
  Assessed using the Central Sensitization Inventory (Total score range from 0 to 100 and higher scores are indicative of a higher degree of symptomatology associated with central sensitization)
Central Sensitization | 6 months
  Assessed using the Central Sensitization Inventory (Total score range from 0 to 100 and higher scores are indicative of a higher degree of symptomatology associated with central sensitization)
Knowledge of pain neuroscience | Baseline
  Assessed using the Pain Neurophysiology Questionnaire (Total score range from 0-19 and higher values are indicative of more knowledge on pain neurophysiology)
Knowledge of pain neuroscience | 8 weeks
  Assessed using the Pain Neurophysiology Questionnaire (Total score range from 0-19 and higher values are indicative of more knowledge on pain neurophysiology)
Knowledge of pain neuroscience | 6 months
  Assessed using the Pain Neurophysiology Questionnaire (Total score range from 0-19 and higher values are indicative of more knowledge on pain neurophysiology)
Muscular resistance of the deep flexor muscles of the cervical | Baseline
  Assessed using the Deep Neck Flexor Endurance Test (the time, in seconds, that each participant will performed the test position will be recorded)
Muscular resistance of the deep flexor muscles of the cervical | 8 weeks
  Assessed using the Deep Neck Flexor Endurance Test (the time, in seconds, that each participant will performed the test position will be recorded)
Muscular resistance of the deep flexor muscles of the cervical | 6 months
  Assessed using the Deep Neck Flexor Endurance Test (the time, in seconds, that each participant will performed the test position will be recorded)
Muscular endurance of the deep cervical extensor muscles | Baseline
  Assessed using the Cervical Extensor Endurance Test (the time, in seconds, that each participant will performed the test position will be recorded)
Muscular endurance of the deep cervical extensor muscles | 8 weeks
  Assessed using the Cervical Extensor Endurance Test (the time, in seconds, that each participant will performed the test position will be recorded)
Muscular endurance of the deep cervical extensor muscles | 6 months
  Assessed using the Cervical Extensor Endurance Test (the time, in seconds, that each participant will performed the test position will be recorded)
Muscular resistance of the stabilizing muscles of the scapular girdle | Baseline
  Assessed using the Scapular Muscle Endurance Test (the time, in seconds, that each participant will performed the test position will be recorded)
Muscular resistance of the stabilizing muscles of the scapular girdle | 8 weeks
  Assessed using the Scapular Muscle Endurance Test (the time, in seconds, that each participant will performed the test position will be recorded)
Muscular resistance of the stabilizing muscles of the scapular girdle | 6 months
  Assessed using the Scapular Muscle Endurance Test (the time, in seconds, that each participant will performed the test position will be recorded)
Pressure Pain Threshold | Baseline
  Assessed using the algometer (the point of minimum pressure that induces a pain sensation will be recorded)
Pressure Pain Threshold | 8 weeks
  Assessed using the algometer (the point of minimum pressure that induces a pain sensation will be recorded)
Pressure Pain Threshold | 6 months
  Assessed using the algometer (the point of minimum pressure that induces a pain sensation will be recorded)

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Andias, MD, Principal Investigator — University of Aveiro
Locations (3):
- Portugal (3):
  - Adolfo Portela High School, Aveiro
  - Dr. Jaime Magalhães Lima High School, Aveiro
  - José Estevão High School, Aveiro

IPD SHARING:
Plan to Share IPD: No